CLINICAL TRIAL: NCT07091461
Title: HOMe-IMprove Telerrehabilitation System for CHilDren With Cerebral Palsy
Brief Title: HOMe-IMprove Telerrehabilitation System
Acronym: HOMIMTES-CHilD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOMIMTES-CHilD
Record Dates: First submitted 2025-07-07; First posted 2025-07-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cerebral Palsy Infantile
Keywords: home; children; infantile cerebral palsy; family; upper extremity; balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOME Kit Tablet Telerehabilitation (Experimental): Participants in this arm will receive a structured telerehabilitation program using the HOME Kit Tablet system, which includes a touchscreen tablet with therapeutic software, inertial measurement unit (IMU) sensors, digital scales, a K-wand, and a stabilometric platform. Sessions are remotely supervised in real time by a trained physiotherapist who personalizes the activity protocol according to individual performance.
  Interventions: Device: HOME Kit Tablet-based Telerehabilitation
- Conventional Home Physiotherapy (Active Comparator): Participants in this arm will follow a conventional home rehabilitation protocol, focusing on upper limb function and postural control. The protocol includes traditional exercises prescribed and explained by a physiotherapist. Follow-up will be conducted through weekly phone calls to reinforce adherence and resolve concerns.
  Interventions: Other: Conventional Home Physiotherapy

INTERVENTIONS:
Device: HOME Kit Tablet-based Telerehabilitation — Device-based behavioral intervention (motor, cognitive, and communication rehabilitation)
  Arms: HOME Kit Tablet Telerehabilitation
Other: Conventional Home Physiotherapy — Participants in this arm will follow a conventional home rehabilitation protocol, focusing on upper limb function and postural control. The protocol includes traditional exercises prescribed and explained by a physiotherapist. Follow-up will be conducted through weekly phone calls to reinforce adherence and resolve concerns.
  Arms: Conventional Home Physiotherapy

SUMMARY:
This pilot study aims to assess the feasibility, adherence, and preliminary efficacy of a home-based telerehabilitation protocol using the HOME Kit Tablet system in children aged 6 to 18 years with cerebral palsy. The study follows a randomized controlled design with parallel groups and single-blind evaluation. The intervention group will use a digitally supervised rehabilitation system, while the control group will follow a traditional home therapy protocol without technological tools.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of infantile unilateral cerebral palsy
* Age between 6 and 18 years
* Stable home Wi-Fi access and space to perform exercises
* Manual Ability Classification System (MACS) level ≤ 3
* Informed consent from legal guardian and assent from the child (if <12 years)

Exclusion Criteria:

* Severe neurological or psychiatric comorbidities
* Recent orthopedic surgery (<12 months) or botulinum toxin treatment (<6 months)
* Concurrent participation in other intervention studies

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in postural control assessed by stabilometric platform | baseline, immediately after the intervention, 1 month after intervention
  Postural control is evaluated using a stabilometric platform, which quantitatively measures center of pressure (CoP) displacement and sway area during quiet standing. The main outcome is the mean sway area in square centimeters (cm²), with lower values indicating better postural stability.
Change in balance performance assessed by the Pediatric Berg Balance Scale (PBS) | baseline, immediately after the intervention, 1 month after intervention
  The PBS is a 14-item observational tool designed to measure balance in children. Scores range from 0 to 56; higher scores indicate better balance function.
Change in unimanual hand function assessed by the Assisting Hand Assessment (AHA) | baseline, immediately after the intervention, 1 month after intervention
  The AHA measures how effectively children with unilateral cerebral palsy use their affected hand in bimanual tasks. Total scores range from 0 to 100; higher scores indicate better hand function.
Change in upper limb performance assessed by the Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) | baseline, immediately after the intervention, 1 month after intervention
  The SHUEE evaluates spontaneous and dynamic use of the upper limb. Scores range from 0 to 100; higher scores indicate better function.
Change in manual ability assessed by the Children's Hand-use Experience Questionnaire (CHEQ) | baseline, immediately after the intervention, 1 month after intervention
  The CHEQ is a parent-reported measure that assesses the child's experience using their affected hand in daily tasks. Item scores and mean summary scores; higher scores reflect better experiences.
Change in gross manual dexterity assessed by the Box and Block Test | baseline, immediately after the intervention, 1 month after intervention
  The Box and Block Test assesses gross manual dexterity by counting the number of blocks moved from one compartment to another in one minute. Higher numbers indicate better manual dexterity.

SECONDARY OUTCOMES:
Change in participation in daily activities assessed by the Participation and Environment Measure for Children and Youth (PEM-CY) | baseline, immediately after the intervention, 1 month after intervention
  The PEM-CY questionnaire evaluates participation frequency, involvement, and environmental supports and barriers across home, school, and community settings in children and youth. Scores are reported as frequency (number of activities per week), level of involvement (1-5 scale), and percentage of environmental barriers identified. Higher scores in frequency and involvement indicate greater participation, while higher percentages of environmental barriers reflect more challenges. Outcomes will be summarized for each domain (home, school, community) separately.
Change in individual goal achievement assessed by Goal Attainment Scaling (GAS) | baseline, immediately after the intervention
  Goal Attainment Scaling (GAS) is a participant-centered outcome measure that evaluates the extent to which individualized rehabilitation goals are achieved. Each participant collaborates with the therapist to set specific goals at baseline, which are rated on a 5-point scale ranging from -2 (much less than expected outcome) to +2 (much more than expected outcome), with 0 representing the expected level of achievement. Higher total GAS scores reflect greater goal attainment and better functional improvement.
Change in occupational performance and satisfaction assessed by the Canadian Occupational Performance Measure (COPM) | baseline, immediately after the intervention, 1 month after intervention
  The COPM measures self-perceived performance and satisfaction in daily activities identified as important by the participant or caregiver. Participants rate their performance and satisfaction on a 10-point scale (1-10), with higher scores indicating better performance and greater satisfaction. The primary outcomes are changes in COPM performance and satisfaction scores between baseline and post-intervention assessments.
Change in user satisfaction evaluated with a 5-point Likert-scale questionnaire | immediately after the intervention.
  User satisfaction with the intervention will be assessed using a structured questionnaire based on a 5-point Likert scale, ranging from 1 (very dissatisfied) to 5 (very satisfied). The total score will be calculated as the mean of individual item responses. Higher scores indicate greater satisfaction with the rehabilitation protocol and the HOME Kit system. The questionnaire includes items related to usability, comfort, perceived usefulness, and motivation.